CLINICAL TRIAL: NCT01218269
Title: A Prospective Evaluation of U-clips for Arterial Microvascular Anastomoses
Brief Title: U-clip Pilot Study in Plastic Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Scott and White Hospital & Clinic (Other)
Responsible Party: Raman Chaos Mahabir, MD, MSc, FRCSC, Scott and White
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SWHospital - 90415
Record Dates: First submitted 2010-10-07; First posted 2010-10-11 (Estimated); Last update posted 2011-03-01 (Estimated); Status verified 2010-09

CONDITIONS: Microvascular Anastomoses
Keywords: anastomoses

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- no arms (Other): all patients will receive the treatment - there is only one arms
  Interventions: Device: nitinol u-clip

INTERVENTIONS:
Device: nitinol u-clip — The U-clip is comprised of nitinol, an alloy of nickel and titanium.
  Other Names: Coalescent Surgical U-CLIPTbl

SUMMARY:
This study will assess the nitinol U-clip as an alternative to conventional microsurgical suture for arterial anastomoses in free tissue transfer.

DETAILED DESCRIPTION:
Within Scott & White, a total of 25 free flaps will be performed using U-clips for microvascular anastomoses in lieu of traditional suturing techniques. Each of these free flaps may be in individual patients or two anastomoses may be included in one patient. Historical controls will be used for comparison of complication rates of U-clip versus sutured anastomoses. Postoperatively, the study participants will be evaluated at 2 weeks (+/- 1 week) and at 3 months (+/- 1 month) follow up.

ELIGIBILITY:
Inclusion Criteria:

* either gender
* any ethnicity
* patient requiring free tissue transfer for complex wound coverage or reconstruction
* patient having arterial anastomotic diameter of at least 2 mm
* patient capable of giving informed consent

Exclusion Criteria:

* less than 18 years of age
* allergy to nitinol or any of its components (nickel or titanium)
* pregnancy
* known coagulopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2009-10; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Flap failure rate compared to published rate for conventional suture anastomoses | will be measured 3 months postoperative (+/- 2 weeks)

SECONDARY OUTCOMES:
Rapid, reproducible, sutureless microvascular arterial anastomoses in free flaps without compromising patient outcomes. | data collected at 3 months postoperative (+/- 2 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Raman C Mahabir, MD, Principal Investigator — Scott & White
Locations (1):
- Scott and White Hospital and Clinic, Temple, Texas, United States